CLINICAL TRIAL: NCT01044316
Title: A Phase III Observer-Blind, Randomized, Controlled, Single-Coordinating Center Pediatric Study in China Comparing Two Doses of a Monovalent Glycoprotein-Conjugated (Diptheria Toxin -CRM197) Vaccine Versus a Tetanus Toxoid-Conjugated Vaccine Using a Local Dosing Regimen in Infants
Brief Title: Study in Infants (6-12 Months) Comparing Two Doses of a Monovalent Glycoprotein-Conjugated (Diptheria Toxin -CRM197) Vaccine Versus a Tetanus Toxoid-Conjugated Vaccine Available for the Prevention of Haemophilus Influenzae Type b Infections in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V37_07
Record Dates: First submitted 2010-01-03; First posted 2010-01-07 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Haemophilus Influenzae Type b (Hib) Infection
Keywords: Haemophilus influenzae type b (Hib); Vaccine; Booster
MeSH Terms: conditions — Haemophilus Infections; Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Biological: Haemophilus influenzae type b (Hib) vaccine
- Arm 2 (Active Comparator)
  Interventions: Biological: Haemophilus influenzae type b (Hib) vaccine

INTERVENTIONS:
Biological: Haemophilus influenzae type b (Hib) vaccine — Comparator study of two commercially available Haemophilus influenzae type b (Hib) vaccines - a monovalent glycoprotein-conjugated (diptheria toxin - CRM197) vaccine and a tetanus toxoid-conjugated vaccine.

SUMMARY:
This study will evaluate the safety and efficacy of two doses of two commercially available vaccines used to prevent Haemophilus influenzae type b infections in children 6-12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants 6-12 months of age.

Exclusion Criteria:

* Prior Hib vaccine administration.
* History of serious reaction(s) following vaccination.
* Any vaccination within 14 days of study vaccination.
* Known or suspected immune impairment.
* For additional entry criteria please refer to the protocol.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 670 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Anti-PRP antibody levels at day 31 post last vaccination | 30 days after last vaccination

SECONDARY OUTCOMES:
Solicited local and systemic reactions, AEs, and SAEs | 30 days post last vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Province, China

REFERENCES:
- [Derived] Jun L, Yuguo C, Zhiguo W, Jinfeng L, Huawei M, Xiuhua L, Yonggui Z, Yanhua X, Kong Y, Hongtao L, Yuliang Z. Assessment of immunogenicity and safety following primary and booster immunisation with a CRM197 -conjugated Haemophilus influenzae type B vaccine in healthy Chinese infants. Int J Clin Pract. 2013 Oct;67(10):971-8. doi: 10.1111/ijcp.12267. Epub 2013 Aug 22. PMID 23964690